CLINICAL TRIAL: NCT02526862
Title: Prevention of Pressure Ulcers in Patients Under Non-Invasive Mechanical Ventilation. Randomized Clinical Trial
Brief Title: Prevention of Pressure Ulcers in Patients Under Non-Invasive Mechanical Ventilation
Acronym: PUPPVMNI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Medical SA (Industry)
Collaborators: Instituto de Investigación Sanitaria Gregorio Marañón (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, David Peña Otero, Nurse, Master of Science, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUPPVMNI_200910
Record Dates: First submitted 2015-08-06; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Failure
Keywords: noninvasive mechanical ventilation (NIVM); continuous positive airway pressure (CPAP) ventilation; bilevel positive airway pressure (BIPAP) ventilation; pressure ulcer (PU); nursing assessment
MeSH Terms: conditions — Respiratory Insufficiency; Microcephaly, Primary Autosomal Recessive, 6; Respiratory Aspiration; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A-Mask or direct interface (No Intervention): Mask or direct interface
- B-Autoadhesive polyurethane dressing (Active Comparator): Protection of the dermis with autoadhesive polyurethane dressing (Allevyn Thin®). The dressing will be standardized cut to avoid bias. The edges shape will be circular. They will be set in nasal bridge and cheekbones, avoiding frontal level. It will be checked every six hours, and if not properly fixed it will be applied again in the same way.
  Interventions: Device: Allevyn Thin®
- C-Semi-permeable hydrogel-foam (Active Comparator): Protection of the dermis with semi-permeable hydrogel-foams adhesive dressing (Askina Transorbent Border®). The dressing will be standardized cut to avoid bias. The edges shape will be circular. They will be set in nasal bridge and cheekbones, avoiding frontal level. It will be checked every six hours, and if not properly fixed it will be applied again in the same way.
  Interventions: Device: Askina Transorbent Border®
- D-Hyper hydrogenated fatty acids (Active Comparator): Protection of the dermis with hyper hydrogenated fatty acids (Linovera®) in the contact areas with the NIVM interface or mask. It will apply with its doser and gently massaged in chin, cheekbones, nasal and frontal bridge as indicated in the product. It will be checked every six hours for proper hydration and if needed it will be applied again in the same way.
  Interventions: Device: Linovera®

INTERVENTIONS:
Device: Allevyn Thin® — Protection of the dermis with autoadhesive polyurethane dressing. The dressing will be standardized cut to avoid bias. The edges shape will be circular. They will be set in nasal bridge and cheekbones, avoiding frontal level. It will be checked every six hours, and if not properly fixed it will be applied again in the same way.
  Arms: B-Autoadhesive polyurethane dressing
Device: Askina Transorbent Border® — Protection of the dermis with semi-permeable hydrogel-foams adhesive dressing. The dressing will be standardized cut to avoid bias. The edges shape will be circular. They will be set in nasal bridge and cheekbones, avoiding frontal level. It will be checked every six hours, and if not properly fixed it will be applied again in the same way.
  Arms: C-Semi-permeable hydrogel-foam
Device: Linovera® — Protection of the dermis with hyper hydrogenated fatty acids. It will be applied with its doser and gently massaged in chin, cheekbones, nasal and frontal bridge as indicated in the product. It will be checked every six hours for proper hydration and if needed it will be applied again in the same way.
  Arms: D-Hyper hydrogenated fatty acids

SUMMARY:
This study aims to test direct application of the Non-Invasive Mechanical Ventilation -NIVM- mask or interface as the most efficient intervention to prevent Pressure Ulcers (PU), compared with other three usual preventive measures which consist in the use of three different medical devices.

DETAILED DESCRIPTION:
Non-Invasive Mechanical Ventilation (NIVM) has turned into a standard in the care of patients with acute respiratory failure. Defined as a support modality to the patient's spontaneous ventilation, it does not use invasive techniques to ventilate, working as an external device named interface or mask, avoiding so the complications associated to the invasive ventilation.

NIVM had been restricted to ICU and Pneumology services, but in the last years it has been extended to ER with good results and it is being also used in the pre-hospital attention and in the home care of chronic patient.

Often, the preferred interface is the oronasal, worst tolerated but associated to best treatment of the acute pathology. In most cases to avoid air leaks, its proper placement generates high pressure on the skin, being able to harm patient's tissues, so that this therapy as intervention for the acute patient has pressure ulcers -PU- as main iatrogenic effect - although 95% of the PU are considered as preventable-.

To diminish the pressure of the mask on the points of the face, nurses protect the most exposed zones with dressings of hydrogel-foam, polyurethane and/or hyperoxygenated fatty acids, trying to prevent PU.

Reviewed studies present a big variability in these practices as well as high dispersion of the results achieved.

Preventive measures are different and even none, as applying the mask or the interface directly could be the most effective treatment in the prevention of PU, avoiding not justified increase of fungible and other resources consumption.

The aim of this study is to test direct application of the mask or interface, as the most efficient intervention, compared with other three usual preventive measures which consist in the use of three different medical devices: autoadhesive polyurethane dressing (Allevyn Thin®), semi-permeable hydrogel-foams adhesive dressing (Askina Transorbent Border®) or hyperoxygenated fatty acids (Linovera®)

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Not tissue injury in face.
* Not structural deformation of the facial anatomy.

Exclusion Criteria:

* Rejects Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Incidence of PU for each group (mean, standard deviation and quartiles) | First 24 hours after the withdrawal of the treatment
  Compare the efficacy of the preventive treatments A, B, C and D - previously described-(meaning by efficacy the no occurrence of PU).
  For definition of PU investigators use the one of the "National Group for the Study and Advice in Pressure Ulcer and Chronic Wounds" (GNEAUPP)

SECONDARY OUTCOMES:
Incidence of total NIVM related PU, by observation registers. | 24 hours after the withdrawal of the treatment
  Total incidence of NIVM related PU within the first 24 hours after the withdrawal of the treatment, registered for the different preventive procedures.
Efficiency of preventive measures for PU related to NIVM, by registering incidence and resources invested -time in hours and consumables in euros- (mean, standard deviation and quartiles for each group) | 24 hours after the withdrawal of the treatment
  Compare the efficacy and efficiency (cost related efficacy) of the preventive treatments A, B, C and D - previously described

CONTACTS AND LOCATIONS:
Overall Officials: David Peña-Otero, M.Sc., Principal Investigator — Nurse. Emergency and Critical Care. Hospital General Universitario Gregorio Marañón. Nursing Faculty. Universidad Rey Juan Carlos. Instituto de Investigación Sanitaria Gregorio Marañón (IiSGM)
Locations (1):
- Emergency and Critical Care. Hospital General Universitario Gregorio Marañón., Madrid, Madrid, Spain